CLINICAL TRIAL: NCT01302028
Title: An Open-label, Parallel Group Study to Assess the Effect of Different Grades of Renal Impairment in Patients With Type 2 Diabetes Mellitus on the Pharmacokinetics, Pharmacodynamics and Safety & Tolerability of ASP1941 Relative to Type 2 Diabetes Mellitus With Normal Renal Function and Healthy Volunteers
Brief Title: Renal Impairment Study With ASP1941
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1941-CL-0064; 2009-011320-61 (EudraCT Number)
Record Dates: First submitted 2011-02-21; First posted 2011-02-23 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Renal Impairment; ASP1941; Pharmacokinetics
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency | interventions — ipragliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Healthy volunteers with normal renal function (Active Comparator): Oral
  Interventions: Drug: ASP1941
- T2DM patient with normal renal function (Experimental): Oral
  Interventions: Drug: ASP1941
- T2DM patient with mild renal impairment (Experimental): Oral
  Interventions: Drug: ASP1941
- T2DM patient with moderate renal impairment (Experimental): Oral
  Interventions: Drug: ASP1941
- T2DM patient with severe renal impairment (Experimental): Oral
  Interventions: Drug: ASP1941

INTERVENTIONS:
Drug: ASP1941 — Oral

SUMMARY:
A study to investigate if the pharmacokinetics of ASP1941 is different in Type 2 Diabetes Mellitus (T2DM) patients with different grades of renal failure compared with T2DM patients with normal renal function and healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Patient with stable type 2 diabetes mellitus or healthy subject
* Subject must have pre-dose estimated Glomerular filtration rate (GFR) values (Modification of diet in renal disease (MDRD) method) at screening of:

  * >90 (normal renal function)
  * 60-90 (mild renal impairment)
  * 30-60 (moderate renal impairment)
  * 15-30 (severe renal impairment)
* BMI between 25.0-40.0 kg/m2, inclusive
* Fasted plasma glucose (FPG) <11.5 mmol/l (type 2 DM patients) or >5.6 mmol/l (Healthy volunteers)

Exclusion Criteria:

* Patients with Type 1 diabetes
* Pulse <40 or >90; SBP >160 mmHg; DBP > 100 mmHg
* T2DM patients who are not on a stable regimen for their current medication (1 month or 5 half lives, whichever is longer) to control their disease
* Healthy Volunteers: Any of the liver function tests above the upper limit of normal
* T2DM: The liver function tests should be within the following ranges:

  * AST/ALT: <2 x ULN
  * Bilirubin: <1.5 x ULN
  * Alk Phos: < 1.5 x ULN
* Patients with renal impairment who have a history of a clinically significant illness (other than renal diseases and T2DM and associated clinical symptoms), medical condition, or laboratory abnormality within 3 months prior to screening
* Patients with renal impairment who have not been on a stable dose of concomitant medications for at least 2 weeks for at least 2 weeks (or 5 halflives, whichever is longer) and/or for whom dose changes are likely to occur during the study
* Patients with T2DM treated with a diet only
* T2DM patients with recent evidence (e.g within the last 6 months) of severe hypoglycemia, for example plasma glucose < 3mmol/l (<55 mg/dl), help from others to resolve the hypo or requiring hospitalization
* T2DM patients with a Hemoglobin value < 9 g/dl (5.6 mmol/l)

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-01-22 (Actual); Primary Completion 2010-06-26 (Actual); Study Completion 2010-06-26 (Actual)

PRIMARY OUTCOMES:
Effect of grade of renal impairment on the pharmacokinetics of ASP1941 | 5 days

SECONDARY OUTCOMES:
Effect of grade of renal impairment on the pharmacodynamics of ASP1941 | 5 days
Assessment of safety through evaluation of adverse events, physical examination, vital sins, lab-tests and 12-lead ECG | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma Europe B.V.
Locations (5):
- Czechia (2):
  - Brno
  - Prague
- Balatonfüred, Hungary
- Warsaw, Poland
- Bratislava, Slovakia

REFERENCES:
- [Derived] Ferrannini E, Veltkamp SA, Smulders RA, Kadokura T. Renal glucose handling: impact of chronic kidney disease and sodium-glucose cotransporter 2 inhibition in patients with type 2 diabetes. Diabetes Care. 2013 May;36(5):1260-5. doi: 10.2337/dc12-1503. Epub 2013 Jan 28. PMID 23359360
- See also: Link to results on Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/study.aspx?ID=6